CLINICAL TRIAL: NCT05369078
Title: Phase I Clinical Study to Evaluate the Safety, Tolerance and Pharmacokinetics of THR-1442 in Chinese Healthy Subjects
Brief Title: Safety, Tolerance and Pharmacokinetics of THR-1442 in Chinese Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newsoara Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Newsoara HYK Biopharmaceutical (Shanghai) Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THR-1442-C-607 （CHN）
Record Dates: First submitted 2021-12-06; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2021-12

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Study includes 2 parts: Single does part and multiple dose part. Single does part and multiple dose part are started same time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THR-1442 20mg Single dose group (Experimental): THR-1442 20mg Single dose group: subject will be administrated 1 dose of 20mg THR-1442 on day1, the follow up till day 7.
  Interventions: Drug: THR-1442 20mg Single dose
- THR-1442 20mg Multiple dose group (Experimental): THR-1442 20mg Multiple dose group: subject will be administrated THR-1442 20mg QD on Day1-Day7, the follow up till day 14.
  Interventions: Drug: THR-1442 20mg Multiple dose group

INTERVENTIONS:
Drug: THR-1442 20mg Single dose — THR-1442 20mg is administrated 1 dose on Day 1, then follow till day 7.
  Arms: THR-1442 20mg Single dose group
Drug: THR-1442 20mg Multiple dose group — THR-1442 20mg is administrated QD for 7days, then follow till day 14.
  Arms: THR-1442 20mg Multiple dose group

SUMMARY:
The purpose of this study was to investigate Safety, tolerability and pharmacokinetics in Chinese healthy subjects.

DETAILED DESCRIPTION:
This was a single center, Phase 1, open-label SAD and MAD study designed to assess safety, tolerability and PK of orally administered THR-1442 tablets in Chinese healthy adults.

Subjects were enrolled to receive 20mg THR-1442 tablet in Single dose group (20mg*1 day) and multiple dose group(20mg*7days).

Blood samples for THR-1442 plasma concentrations were collected 0h till to 48hours.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand and be willing to sign informed consent and voluntarily participate in the study;
2. Chinese women or men aged 18-45 (including 18 and 45) at the time of screening;
3. Men or women who agree to effective contraception from the screening period until 30 days after the last dose in the trial; Agree to take at least one effective contraceptive measure;
4. During screening and baseline, male weight ≥ 50.0kg, female weight ≥ 45.0kg, body mass index (BMI) in the range of 19 ~ 25.0kg/m2 (including 19 and 25.0kg/m2), [BMI = weight (kg) / height 2 (M2)];

Exclusion Criteria:

1. According to the judgment of the site investigators, including clinical significant medical history in CNS, CV system, respiratory system, blood / hematopoietic system, gastrointestinal system, liver / kidney system，etc;
2. Subjects with specific allergic history or allergic constitution such as drugs, food and pollen, or allergic to SGLT2 inhibitors or similar drugs;
3. Alcoholics (drinking 14 units per week, each unit equivalent to 360mL beer or 150mL wine or 45mL alcohol of 40% alcohol), drug or drug dependence subjects; Smokers (smoking > 5 cigarettes per day or the same amount of other tobacco products);
4. Subjects with a history of bladder dysfunction, such as urinary incontinence, frequent urination or nocturia;
5. Blood donation within 3 months before screening, including component blood or massive blood loss (≥ 200ml), receiving blood transfusion or using blood products;
6. Subjects who used prescription drugs, traditional Chinese medicine, over-the-counter drugs (OTC), vitamins, dietary supplements or supplements (e.g. ginseng) within 4 weeks before the first administration;
7. From 7 days before the first dose to the whole study period, subjects who are unwilling or unable to guarantee to forbid by the following: no smoking, no alcohol, no caffeine containing products (including chocolate, tea, coffee, cola, etc.) and avoid strenuous exercise;
8. Those who are unwilling or unable to guarantee to forbid pitaya, grapefruit, mango, carambola, fruit juice and spicy food containing the above fruits from 7 days before taking the medicine and the whole test period;
9. The subject was unable to swallow the study drug or had gastrointestinal diseases leading to absorption disorders;
10. Subjects who had participated in any drug or medical device clinical trial within 3 months before screening;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Collect and evaluate TEAEs (including clinical AEs and Lab AEs) of THR-1442 in healthy subjects during study | Single dose：Baseline to day 7 ； Multiple dose：Baseline to Day14
  Collect data(TEAEs including clinical AEs and lab AEs) on Day7 and Day14 to evaluate THR1442 safety and tolerability

SECONDARY OUTCOMES:
Select and evaluate pharmacokinetic characteristics(AUC) of THR-1442 in healthy subjects during the study | Single dose：Day1-Day7； Multiple dose：Day1- Day14
  Collect blood samples on Single dose part and multiple dose part to evaluate THR1442 PK parameters （AUC）
Select and evaluate pharmacokinetic characteristics(Cmax) of THR-1442 in healthy subjects during the study | Single dose：Day1-Day7； Multiple dose：Day1- Day14
  Collect blood samples on Single dose part and multiple dose part to evaluate THR1442 PK parameters （Cmax）

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's hospital, Hangzhou, Zhejiang, China